CLINICAL TRIAL: NCT04625920
Title: A Virtual Reality System for Pain and Anxiety Management During Outpatient Hysteroscopy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tel-Aviv Sourasky Medical Center (Other Government)
Responsible Party: Principal Investigator, michal roll, Director, Head of Clinical Trails Department, Principal Investigator, Clinical Professor, Tel-Aviv Sourasky Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 0793-19
Record Dates: First submitted 2020-10-27; First posted 2020-11-12 (Actual); Last update posted 2020-11-12 (Actual); Status verified 2020-11

CONDITIONS: Infertility; Vaginal Blood Loss
Keywords: Hysteroscopy; VR; Vurtual reality
MeSH Terms: conditions — Infertility; Uterine Hemorrhage

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Virtual reality (Experimental): women allocated to undergo hysteroscopy with Vr System
  Interventions: Device: SootheVR: AppliedVR, Los Angeles, California
- Standart care (Experimental): women allocated to undergo hysteroscopy without VR
  Interventions: Device: SootheVR: AppliedVR, Los Angeles, California

INTERVENTIONS:
Device: SootheVR: AppliedVR, Los Angeles, California — a head-mounted display

SUMMARY:
To evaluate the effectiveness of VR as a distraction technique in the management of acute pain and anxiety during operative hysteroscopy in the outpatient setting.

DETAILED DESCRIPTION:
A prospective, open-label, randomized control trial in a tertiary university-affiliated medical center between April to August 2020. Overall, 100 women will be randomly allocated to undergo operative hysteroscopy either with the use of VR (study group) or with standard treatment (control group). The primary outcome measures includ self-reported pain, anxiety scores, and vital parameters as pulse rate (PR) and respiratory rate (RR). Pain and anxiety outcomes were measured as numeric rating scores.

ELIGIBILITY:
Inclusion Criteria:

* . Women with suspected infection
* women considered not suitable to undergo an office hysteroscopy
* women who reported the use of analgesia 6 hours prior to the procedure.

Exclusion Criteria:

* patient needed office hysteroscopy

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 100 (Actual)
Dates: Start 2020-04-10 (Actual); Primary Completion 2020-09-20 (Actual); Study Completion 2020-09-30 (Actual)

PRIMARY OUTCOMES:
Assessments of pain through physiological parameters | 10 minutes
  Assessments of pain through physiological parameters of pulse rate. Heart Rate will be measured using Heart Rate-beats per minute.
Assessments of pain through pain score parameter | 10 minutes
  Assessments of pain through pain score parameter of the NRS questionnaire. Pain will be measured using the Numeric Rating Scale (NRS) which is a 11 point scale from 0 to 10 which is a validated score of measuring pain and anxiety in which 0 is no pain and 10 is the worst imaginable pain and or anxiety.

CONTACTS AND LOCATIONS:
Overall Officials: eli shprecher, Prof, Study Chair — souraski MC
Locations (2):
- Israel (2):
  - Lis Maternity Hospital, Tel Aviv Sourasky Medical Center, Tel Aviv
  - Souraski MC, Tel Aviv

IPD SHARING:
Plan to Share IPD: No